CLINICAL TRIAL: NCT02495558
Title: Pilot Study of the Cough Reflex Assessment in Patients With Tracheostomy Cannula Following Severe Acquired Brain Injury
Brief Title: Cough Assessment in Patients With Severe Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Irene Battel, Speech and Language Therapist, IRCCS San Camillo, Venezia, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TRGCA
Record Dates: First submitted 2015-07-02; First posted 2015-07-13 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Tracheostomy Complication; Acquired Brain Injury; Brain Injury; Pneumonia
Keywords: Cough Reflex test; Decannulation
MeSH Terms: conditions — Brain Injuries; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Tracheostomy (Experimental): Assessment of reflex cough Assessment of the deccanultation outcome (follow-up)
  Interventions: Other: Reflex Cough Test

INTERVENTIONS:
Other: Reflex Cough Test — Peak of Cough Expiratory Flow of the reflex cough

SUMMARY:
The cough assessment is fundamental in the weaning process as it gives information on the possibility to expel food and secretion out from the airways. The majority of persons suffering from severe acquired brain injury are not able to cough voluntary due to severe cognitive deficit. In the present study, it would be evaluated the intensity of the reflex cough (RC) and the results would be correlated with weaning outcome.

DETAILED DESCRIPTION:
All the participants will undergo firstly to the RC assessment. RC would be trigged by the inhalation of 0.4M of citric acid solution using the ultrasonic nebulizer (MO-03 Norditalia Elettromedicali). The face mask would be connected with the spirometer and the nebulizer via a bidirectional valve in order to measure Peak of Cough Expiratory Flow (PCEF) of the RC. Secondly, it would be assessed parameters of the weaning protocol in order to verify the feasible of removing the tracheostomy cannula. Hence, if the previous assessments are positive, the cannula 's patients would be removed. The follow-up would be taken after 96 hours from the decannulation in order to verify the outcome of weaning.

In this study, it would be recruited a number of 30 consecutive patients admitted to IRCCS Ospedale San Camillo. The data would be firstly analyzed using Kolmogorov-Smirnov test in order to verify the distribution. Secondly it would be chosen to t-test for parametric outcomes or Wilcoxon non parametric outcomes. Thirdly, the correlation between the Peak of Cough Expiratory Flow of the RC and the weaning outcome would be completed using Pearson Test (parametric) or Spearman test (non parametric).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Acquired Brain Injury
* presence of tracheostomy cannula and positive cupping trial
* provide informed consent independently

Exclusion Criteria:

* presence of allergy to citrus;
* presence of asthma
* presence of mechanical ventilation;
* presence of trachomalacia
* presence of laryngeal stenosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
PCEF of the reflex cough | 8 weeks
  Peak of expiratory flow during reflex cough in patients with severe acquired brain injury

SECONDARY OUTCOMES:
PCEF of the reflex cough after decannulation | 9 weeks
  The peak cough expiratory flow would be assessed after 96 hours post decannulation.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Enrichi, Principal Investigator — claudia.enrichi@ospedalesancamillo.net
Locations (1):
- Fondazione Ospedale San Camillo IRCCS, Venice, Venice, Italy

REFERENCES:
- [Background] Bach JR, Saporito LR. Criteria for extubation and tracheostomy tube removal for patients with ventilatory failure. A different approach to weaning. Chest. 1996 Dec;110(6):1566-71. doi: 10.1378/chest.110.6.1566. PMID 8989078
- [Background] Bittner EA, Schmidt UH. The ventilator liberation process: update on technique, timing, and termination of tracheostomy. Respir Care. 2012 Oct;57(10):1626-34. doi: 10.4187/respcare.01914. PMID 23013900
- [Background] McCool FD. Global physiology and pathophysiology of cough: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):48S-53S. doi: 10.1378/chest.129.1_suppl.48S. PMID 16428691
- [Background] Miles A, Huckabee ML. Intra- and inter-rater reliability for judgement of cough following citric acid inhalation. Int J Speech Lang Pathol. 2013 Apr;15(2):209-15. doi: 10.3109/17549507.2012.692812. Epub 2012 Aug 8. PMID 22873621